CLINICAL TRIAL: NCT04569656
Title: Pilot Study for the Evaluation of the Parameters of Activity of a Preparation of PHGG and Sodium Hyaluronate in Chronic Constipation in Patients With Parkinson's Disease
Brief Title: Treatment of Chronic Constipation in Parkinson's Disease
Acronym: PHGG-PD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: IRCCS San Raffaele Roma (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RP 04/15
Record Dates: First submitted 2020-09-24; First posted 2020-09-30 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2022-10

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment (Experimental): 6 week treatment with Stick pack 30 ml containing PHGG 5 gr e Hyaluronic Acid 200 mg
  Interventions: Drug: hydrolyzed guar gum

INTERVENTIONS:
Drug: hydrolyzed guar gum — treatment with Stick pack 30 ml containing PHGG 5 gr e Hyaluronic Acid 200 mg for 6 weeks
  Other Names: PHGG

SUMMARY:
Chronic constipation is the most common gastrointestinal symptom reported by PD patients; it could be one of the manifestations of disease onset.

PHGG fiber is extracted from a herbaceous plant (Cyamopsis Tetra-Gonolobus, family: Leguminosae) of Indian origin: it produces 5/9 pods containing seeds which produce the famous guar gum, that is a natural polysaccharide.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a chronic and progressive neurodegenerative disorder characterized by motor symptoms. In recent years it has become clear that motor symptoms are associated with non-motor and non-dopaminergic symptoms throughout the natural progression of the disease, and sometimes even before the onset of motor manifestations.

Chronic constipation is the most common gastrointestinal symptom reported by PD patients; it could be one of the manifestations of disease onset.

In the past, constipation was considered a side effect of neurological therapy, but more recent studies have evidenced that it is widely present in patients with early untreated PD too and it may precede of years the onset of motor symptoms.

The prevalence of constipation can reach 80% of patients with PD, with an incidence of decreased stool frequency (less than 3 bowel movements per week) of 57-67% of patients.

Although constipation should be interpreted as part of the disease, patients often don't link it to PD, with the result that it may be neglected or poorly managed. Moreover, continuous and incongruous use of laxatives, that are often used in increasing doses in order to maintain efficacy, may cause the onset of abdominal pain and diarrhoea with the risk of bowel incontinence and other side effects.

Constipation also adversely affects quality of life of PD patients: beyond being an annoying symptom, it may also cause other serious gastrointestinal pathologies (i.e. magacolon, intestinal pseudo-obstruction, volvolus, bowel perforation). Moreover, constipation can directly or indirectly influence the absorption of PD drugs, with the result of a poor control on motor symptoms.

Afterwards, finding an effective treatment of constipation would be very important for quality of life of PD patients; this treatment should be easy to be administered and should not have any interference with other PD drugs.

PHGG fiber is extracted from a herbaceous plant (Cyamopsis Tetra-Gonolobus, family: Leguminosae) of Indian origin: it produces 5/9 pods containing seeds which produce the famous guar gum, that is a natural polysaccharide. It differs from fibers derived from other plants for its high content of Galactomannan. Guar gum (referred to as GG) is classified in the European list of additives under the symbol E 412. Recently, a partially hydrolyzed guar gum (indicated with the abbreviation PHGG) has been developed. Unlike the original and other fibers (eg. Psillium), it has the characteristic to remain liquid and, due to its low molecular weight, to not turn into gel. The introduction of molecules of water (hydrolysis), by an enzyme called Mannanase, reduces the length and the molecular weight of guar gum and creates a fiber with unique properties: by remaining liquid, it does not cause bloating, flatulence and meteorism, that are adverse events typically associated to other fibers. The association with sodium hyaluronate (low molecular weight depolymerizes) rapidly attracting water and amplifying the desired clinical effect.

The aim of this pilot research study is to investigate the effectiveness of this formula (Stick pack 30 ml containing PHGG 5 g and Hyaluronic 200 mg) in PD patients affected by constipation.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic PD according to UK PDS Brain Bank Clinical Diagnostic Criteria.
* Chronic constipation according to Roma III criteria for chronic functional constipation lasting from at least 6 months.
* Absence of dementia.
* Patients who are able to understand and sign the informed consent for participation in the study

Exclusion Criteria:

* People who suffer from other comorbidities that could interfere with the results of the study according to the investigator.
* People who are not able to provide reliable answers to the questionnaire according to the opinion of the investigator.
* Inclusion in other clinical trials at the time of the visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2016-02-02 (Actual); Primary Completion 2016-12-20 (Actual); Study Completion 2016-12-20 (Actual)

PRIMARY OUTCOMES:
to investigate the effectiveness of the preparation of PHGG and sodium hyaluronate on symptoms of PD patients with chronic constipation | trough study completation, an average of 6 weeks
  using the scale the Patient Assessment of Constipation-Symptoms PAC-SYM The 12-item questionnaire is divided into three symptom subscales: abdominal (four items); rectal (three items); and stool (five items). Items are scored on 5-point Likert scales, with scores ranging from 0 to 4 (0 = 'symptom absent', 1 = 'mild', 2 = 'moderate', 3 = 'severe' and 4 = 'very severe'). A mean total score in the range of 0-4 is generated by dividing the total score by the number of questions completed; the lower the total score, the lower the symptom burden.
to investigate the effectiveness of the preparation of PHGG and sodium hyaluronate on symptoms of PD patients with chronic constipation | trough study completation, an average of 6 weeks
  Bristol Stool Chart
to investigate the effectiveness of the preparation of PHGG and sodium hyaluronate on quality of life of PD patients with chronic constipation | trough study completation, an average of 6 weeks
  using Patient Assessment of Constipation Quality of Life PAC-QOL subcategorized to 4 items on physical discomfort, 8 items on psychosocial discomfort, 5 items on treatment satisfaction, and finally 11 items on worries and discomfort. Response choice is a Likert scale from 0 to 4. Higher scores mean higher negative effects on quality of life. Items 25, 26, 27, and 28 should be scored reversed because they are positive questions.

SECONDARY OUTCOMES:
To investigate compliance to treatment. | through study completion, an average of 6 weeks
  assessment of compliance by Clinical Global Impression (CGI) for patient, study drug accountability and a questionnaire for compliance.
  comprises two companion one-item measures evaluating the following: (a) severity of psychopathology from 1 to 7 and (b) change from the initiation of treatment on a similar seven-point scale
To investigate acceptance to treatment. | through study completion, an average of 6 weeks
  assessment of acceptance by Clinical Global Impression (CGI) for patient, study drug accountability.
  comprises two companion one-item measures evaluating the following: (a) severity of psychopathology from 1 to 7 and (b) change from the initiation of treatment on a similar seven-point scale
To investigate adherence to treatment. | through study completion, an average of 6 weeks
  assessment of adherence to treatment by Clinical Global Impression (CGI) for patient, study drug accountability.
  comprises two companion one-item measures evaluating the following: (a) severity of psychopathology from 1 to 7 and (b) change from the initiation of treatment on a similar seven-point scale

CONTACTS AND LOCATIONS:
Overall Officials: fabrizio stocchi, md phd, Principal Investigator — IRCCS San Raffaele
Locations (1):
- IRCCS San Raffaele, Roma, Italy

IPD SHARING:
Plan to Share IPD: Yes
after the end of study
Supporting Information: Study Protocol
Time Frame: after the study
Access Criteria: request by email

REFERENCES:
- [Derived] Vacca L, Proietti S, Bravi D, Radicati FG, Stocchi F. Effectiveness of an herbaceous derivatives, PHGG, plus sodium hyaluronate in the treatment of chronic constipation in patients with Parkinson's disease: a pilot study. Neurol Sci. 2022 Feb;43(2):1055-1059. doi: 10.1007/s10072-021-05342-8. Epub 2021 Jun 4. PMID 34086122